CLINICAL TRIAL: NCT04504188
Title: Optimizing Beta Blocker Dosage in Women While Using the Wearable Cardioverter Defibrillator
Acronym: OPT-BB WOMEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90D0229
Record Dates: First submitted 2020-07-31; First posted 2020-08-07 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Cardiomyopathies; Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure

STUDY DESIGN:
Intervention Model Description: Subjects will wear an FDA-approved WCD with a 3 month follow-up period. Heart rate (HR) will be continuously monitored by the WCD. Every two weeks a report showing daily HR trends will be emailed to the healthcare provider. The healthcare provider will also receive a HR control alert if the HR exceeds a predetermined threshold for 3 days in a row.
  Based on this information, clinicians should follow guideline-directed medical therapy (GDMT) to add or titrate medication accordingly. The goal of these changes will be to achieve the average nighttime HR to recommended guidelines (<70 bpm) by the end of WCD use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Heart Rate Monitor Enhanced Treatment Optimization (Experimental): Subjects will wear an FDA-approved WCD with a 3 month follow-up period. Heart rate (HR) will be continuously monitored by the WCD.
  Interventions: Device: Heart Rate Monitor Enhanced Treatment Optimization

INTERVENTIONS:
Device: Heart Rate Monitor Enhanced Treatment Optimization — Heart rate (HR) will be continuously monitored by the WCD. Every two weeks a report showing daily HR trends will be emailed to the healthcare provider. The healthcare provider will also receive a HR control alert if the HR exceeds a predetermined threshold for 3 days in a row.
  Other Names: LifeVest Wearable Cardioverter Defibrillator

SUMMARY:
The primary objective of this pilot study is to document the percentage achievement in effective HR control (average nighttime HR < 70 bpm) during WCD use in a cohort of female patients with cardiomyopathy in an outpatient setting using continuous heart rate (HR) trends data from the WCD to optimize BB/ivabradine dosage, as compared to a prior historical control.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to document the percentage achievement in effective HR control (average nighttime HR < 70 bpm) during WCD use in a cohort of female patients with cardiomyopathy in an outpatient setting using continuous heart rate (HR) trends data from the WCD to optimize BB/ivabradine dosage, as compared to a prior historical control.

Adult female patients (18 years or older) who are prescribed the wearable cardioverter defibrillator (WCD) for 3 months for ischemic or non-ischemic cardiomyopathy with a low ejection fraction.

Subjects will wear an FDA-approved WCD with a 3 month follow-up period. Heart rate (HR) will be continuously monitored by the WCD. Every two weeks a report showing daily HR trends will be emailed to the healthcare provider. The healthcare provider will also receive a HR control alert if the HR exceeds a predetermined threshold for 3 days in a row.

Based on this information, clinicians should follow guideline-directed medical therapy (GDMT) to add or titrate medication accordingly. The goal of these changes will be to achieve the average nighttime HR to recommended guidelines (<70 bpm) by the end of WCD use.

ELIGIBILITY:
Inclusion Criteria for Screening Phase:

* Female patients with newly diagnosed (never hospitalized for HF in the last 30 days prior to enrollment) ischemic or non-ischemic cardiomyopathy and an EF ≤ 35% at the time of WCD prescription.
* Patients prescribed the WCD for an intended 90 ± 14 days of use.
* Patients have used the WCD for no more than 14 days from the day of consent.
* Patients 18 years of age or older at the time of consent.

Inclusion Criteria for Continuation Phase:

-After the first 2 weeks of WCD wear, only actively wearing patients averaging at least 105 hours of WCD wear per week (or 15 hours/day) are eligible to continue.

Exclusion Criteria for Screening Phase:

* Patients with a known contraindication or intolerance to beta-blocker therapy.
* Patients with permanent atrial fibrillation.
* Patients who have a pacemaker.
* Patients with a current or prior implantable cardioverter defibrillator (ICD).
* Patients who are self-reporting to be pregnant.
* Patients with known congenital or inherited heart disease.
* Patients participating in another interventional clinical trial.
* Patients not expected to live longer than 3 months.

Exclusion Criteria for Continuation Phase:

-Patients ending WCD use within the first two weeks of use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Control | 90 days
  The primary objective of this study is to document the percentage achievement in effective HR control (average nighttime HR < 70 bpm) during WCD use in female patients.

SECONDARY OUTCOMES:
Heart Rate Control in Ischemic vs. Non-ischemic Patients | 90 days
  To document the percentage achievement in effective HR control in ischemic vs. non-ischemic patients
Change in Average Nighttime Resting Heart Rate | 90 days
  Change in Average Nighttime Resting Heart Rate Monitored vs. Historic Heart Rate Control over the course of WCD use.
Changes in the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 90 days
  To observe changes in quality of life over the course of WCD use using the KCCQ-12 Questionnaire. Higher scores on the KCCQ reflect better health status (range 0-100)
Changes in (European Quality of Life 5 Dimension Questionnaire (EQ-5D-5L) | 90 days
  To observe changes in quality of life over the course of WCD use using the EQ-5D-5L Questionnaire. Higher scores on the EQ-5D-5L reflect better health status (range 0-100)
Changes in Functional Capacity | 90 days
  To observe changes in functional capacity as measured by average daily step count over the course of WCD use.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD PHD, Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - TriHealth Hatton Research Institute, Cincinnati, Ohio
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - CardioVoyage, McKinney, Texas
  - CAMC, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No